CLINICAL TRIAL: NCT06534684
Title: The Cerebral and Cognitive Changes After Intermittent Theta Burst Stimulation (iTBS) Treatment for Depression A Randomised Double-blind Sham-controlled Trial
Brief Title: The Cerebral and Cognitive Changes After Intermittent Theta Burst Stimulation (iTBS) Treatment for Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of North Norway (Other)
Collaborators: UiT The Arctic University of Norway (Other)
Responsible Party: Principal Investigator, Per Aslaksen, Professor, University Hospital of North Norway
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 715272
Record Dates: First submitted 2024-05-25; First posted 2024-08-02 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Depression, Unipolar; Depression Moderate
MeSH Terms: conditions — Depressive Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intermittent Theta Burst Stimulation (Active Comparator): Stimulation will be performed with a Mag & More PowerMag EEG 100 system with a double PMD70 p-cool (fluid-cooled) figure-of-eight coil.
  Interventions: Device: Intermittent Theta Burst Stimulation
- Sham Intermittent Theta Burst Stimulation (Placebo Comparator): Sham stimulation will be performed by the Mag & More PowerMag EEG 100 system double PMD70 p-cool figure-of-eight coil Sham system.
  Interventions: Device: Intermittent Theta Burst Stimulation

INTERVENTIONS:
Device: Intermittent Theta Burst Stimulation — Intermittent Theta Burst Stimulation will be delivered with 120% of resting motor threshold with triplet 50 Hz bursts repeated at 5 Hz; 2 seconds on and 8 s off, 600 pulses per session with a total duration of 3 min 9 s. Treatment will be provided for 10 days for two consecutive weeks (except Saturdays and Sundays).

SUMMARY:
The present project aims to assess the neurocognitive impact of a two-week once-a-day regimen of intermittent theta burst stimulation (iTBS) compared to sham iTBS, when targeting the left dorsolateral prefrontal cortex (LDLPFC) in clinically depressed outpatients. The study investigates the relationships between changes in cerebral measures and cognitive performance on an N-back task in relation to the antidepressive effect following iTBS.

DETAILED DESCRIPTION:
The study is a randomized sham controlled double blind clinical trial in which the changes in cortical functions associated with the anti-depressive effect of two weeks of once-a-day neuronavigated iTBS over the left dorsolateral prefrontal cortex (LDLPFC) will be investigated in comparison to sham iTBS. Participants will be recruited prospectively, and the study is performed at a single university hospital. After written informed consent is obtained from eligible, volunteering patients, baseline measurements will be administrated, and the patient will be allocated to either sham or active iTBS once a day for 10 consecutive workdays. A total of three measurements will take place, namely at baseline prior to iTBS treatment, after two weeks with iTBS treatment (posttest) and four weeks after (follow-up). The primary outcome measures will be assessed from baseline to the posttest.

ELIGIBILITY:
Inclusion criteria:

* Patients must meet the diagnostic criteria of at least a moderate depression
* The duration of the current depressive episode must have lasted more than 2 weeks but less than 2 years
* Drug therapy must have been stable for the last three weeks prior to the first treatment day with iTBS
* Patients must volunteer to provide informed consent, be able to follow the treatment schedule and have a satisfactory safety screening for iTBS and MRI

Exclusion criteria:

* The current depressive episode is in the mild range
* The current episode fulfills the criteria for a major depressive episode requiring inpatient treatment and/or electroconvulsive therapy,
* The current depressive episode is clearly triggered by grief or a recent major stressful life event
* Bipolar disorder
* Borderline personality disorder
* Psychotic symptoms
* Alcohol or substance abuse/addiction in the last 6 months
* Current eating disorders
* Obsessive- compulsive disorders
* Post-traumatic stress disorder
* A life-time medical history of seizure
* Neurological or neurosurgical pathologies
* Cardiac or systemic disease
* Metallic prosthetic material or foreign objects (pacemakers, prosthetic eye equipment, etc.)
* Autism
* Pregnancy
* Currently using of antipsychotic medication or benzodiazepines - or any medication that interferes with motor threshold excitability

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-02-12 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2029-02-12 (Estimated)

PRIMARY OUTCOMES:
Data from magnetic resonance imaging - white matter integrity | Change from the pretest to the posttest after 10 treatments with iTBS, an average of 15 days
  Differences between groups when comparing intermittent theta burst stimulation versus sham intermittent theta burst stimulation in anatomical measures of cerebral white matter integrity quantified by fractional anisotropy measured by diffusion tensor imaging (DTI) obtained from magnetic resonance imaging (MRI).
Data from magnetic resonance imaging - cortical thickness | Change from the pretest to the posttest after 10 treatments with iTBS, an average of 15 days
  Differences between groups when comparing intermittent theta burst stimulation versus sham intermittent theta burst stimulation in anatomical measures of thickness in cerebral gray matter thickness quantified by T1-weighted magnetic resonance imaging (MRI).
Data from magnetic resonance imaging - cerebral activity | Change from the pretest to the posttest after 10 treatments with iTBS, an average of 15 days
  Differences between groups when comparing intermittent theta burst stimulation versus sham intermittent theta burst stimulation in cerebral activity quantified by blood-oxygen-level-dependent (BOLD) responses measured by functional resonance imaging (fMRI).

SECONDARY OUTCOMES:
Performance on a N-back cognitive test | Change from the pretest to the posttest after 10 treatments with iTBS, an average of 15 days
  Differences between groups when comparing intermittent theta burst stimulation versus sham intermittent theta burst stimulation in behavioral performance on a cognitive task measuring working memory and executive performance when comparing intermittent theta burst stimulation versus sham intermittent theta burst stimulation.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital North Norway, Tromsø, Norway

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data will be made available to other researchers when the study has ended.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be published after completion of the study. The study protocol will be published as soon as possible.

REFERENCES:
- [Derived] Orbo MC, Hoier S, Vangberg TR, Csifcsak G, Gronli OK, Aslaksen PM. The cerebral and cognitive changes after intermittent theta burst stimulation (iTBS) treatment for depression: study protocol for a randomized double-blind sham-controlled trial. Trials. 2024 Nov 11;25(1):752. doi: 10.1186/s13063-024-08606-8. PMID 39529199